CLINICAL TRIAL: NCT06184958
Title: Potential Role of Intravenous Lidocaine Versus Intravenous Ketamine for Pain Management in Fibromyalgia Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, maha sadek El Derh, Assistant professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASUR332/2023
Record Dates: First submitted 2023-12-06; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Anesthesia
Keywords: Fibromyalgia,Ketamine, Lidocaine
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A:Lidocaine group (Active Comparator): 5 mg/Kg lidocaine in 100 ml normal saline given in 40 minutes with 20 minutes follow up to obverse any delayed complication. This procedure will be repeated weekly for 3 weeks
  Interventions: Drug: Lidocaine group
- Group B:Ketamine group (Active Comparator): 0.5 mg/Kg ketamine sulphate in 100 ml normal saline given in 40 minutes with 20 minutes follow up to obverse any delayed complication. This procedure will be repeated weekly for 3 weeks.
  Interventions: Drug: Ketamine group
- Group C:Placebo group (Placebo Comparator): Placebo 100 ml normal saline given in 40 minutes with 20 minutes follow up to obverse any delayed complication. This procedure will be repeated weekly for 3 weeks.
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: Lidocaine group — Group A: Lidocaine group( 25 patients) will receive 5 mg/Kg lidocaine in 100 ml normal saline given in 40 minutes with 20 minutes follow up to obverse any delayed complication. This procedure will be repeated weekly for 3 weeks.
  Arms: Group A:Lidocaine group
Drug: Ketamine group — Group B:Ketamine group(25 patients) will receive 0.5 mg/Kg ketamine sulphate in 100 ml normal saline given in 40 minutes with 20 minutes follow up to obverse any delayed complication. This procedure will be repeated weekly for 3 weeks.
  Arms: Group B:Ketamine group
Drug: Placebo group — Group C:placebo group (25 patients) will receive placebo 100 ml normal saline given in 40 minutes with 20 minutes follow up to obverse any delayed complication. This procedure will be repeated weekly for 3 weeks
  Arms: Group C:Placebo group

SUMMARY:
The aim of the study is to assess the efficacy of intravenous lidocaine versus intravenous ketamine in treatment of fibromyalgia patients.

DETAILED DESCRIPTION:
Adult fibromyalgia patients (25 to 50 years old) suffering from with uncontrolled pain perception will be enrolled although maximum medical treatment is prescribed.

Pre-procedure study tools:

* patients are on regular medical treatment in the form of Cymbalta 60 mg/day, Triptyzol 25 mg/day, and Gabapantin 100 mg/day.
* The following will be done for all the patients:

  1. Full medical history.
  2. Thorough clinical examination.
  3. Visual analogue scale for pain assessment pre and post administration of the study medications.
  4. FM impact Questionnaire (FIQR) for assessment quality of life pre and post administration of the study medications.
  5. ECG.
  6. Laboratory Investigations will include:

Complete blood count (CBC) Erythrocyte sedimentation rate (ESR) with Westergren blot method in (mm) after 1st hour (mm/1st hour).

C-reactive protein (CRP) in (mg/dl) by latex method. Kidney function tests. Liver enzymes. Rheumatoid factor (RF). Anti-nuclear antibody titer (ANA) by indirect immunofluorescence (IIF).

Patients' recruitment, randomization and control of potential bias The sealed, opaque, sequentially-numbered envelopes method for randomization and allocation concealment will used. Identical, opaque, letter-sized envelopes; each containing a white allocation paper (Marked as "Treatment A") will used and a sheet of single-sided carbon paper closest to the front of the envelope (with the carbon side facing the white paper). Finally, the envelopes will be sealed, with signing across the seal. Likewise, another 2 sets will be prepared 25 "Treatment B" envelopes and "Treatment C" envelopes. The three sets (envelopes) will be combined and shuffled thoroughly. Using a pen, marking a number will be done on the front of each envelope sequentially from 1 to 75. Then, will place these envelopes into a plastic container, in numerical order, ready for use.

An investigator (not involved in sequence generation and allocation concealment) will assess patients for eligibility and assigned eligible patients to either lidocaine intravenous infusion (Group A) , ketamine infusion (Group B) or placebo infusion (group C). Participants, care providers, outcomes assessors, and data analysts will be ignorant of the treatment allocation.

All patients will have an intravenous access with a 20G cannula and will be monitored by pulse oximetry, electrocardiogram and non-invasive blood measurement (every 5 minutes). They will be randomly assigned into one of the following three groups:

GROUP A: ( 25 patients) will receive 5 mg/Kg lidocaine in 100 ml normal saline given in 40 minutes with 20 minutes follow up to obverse any delayed complication. This procedure will be repeated weekly for 3 weeks.

GROUP B: ( 25 patients) will receive 0.5 mg/Kg ketamine sulphate in 100 ml normal saline given in 40 minutes with 20 minutes follow up to obverse any delayed complication. This procedure will be repeated weekly for 3 weeks.

Group C: ( 25 patients) will receive placebo 100 ml normal saline given in 40 minutes with 20 minutes follow up to obverse any delayed complication. This procedure will be repeated weekly for 3 weeks.

All patients will be monitored to detect any abnormalities either due to hypersensitivity of the patients or due to potential side effects of lidocaine such as dizziness, fatigue, headache, itchy, warm or red skin, or due to ketamine example hallucination (aborted by 1 mg midazolam), nausea or vomiting, panic attack or memory problems.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FM, diagnosed according to the American College of Rheumatology (ACR) 2016 diagnostic criteria for FM. (Wolfe, F., Clauw, D. J., Fitzcharles, M. A., et al., 2016)

Exclusion Criteria:

* - Known hypersensitivity to any of the given drugs or one of their derivatives (lidocaine or ketamine).
* Known Arrhythmia (Supraventricular or ventricular).
* Pregnant females.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-09-02 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
: Fibromyalgia impact questionnaire with special attention to Visual Analogue Score (VAS). | Assessment will be done weekly for 3 weeks. First assessment will be 1week after first procedure ,on the same day of 2nd injection. 2nd assessment will be on the same day of the 3rd injection . 3rd assessment will be done 1 week after third injection
  Questionnaire to assess degree of pain relieve and improvement of physical activity, a scale from 0-10 where 0 is no pain or limitation and 10 is the worst unbearable pain perception. Asucess is achieved when decline in the scale takes place 3 points out of 10 , where at least reach 5

SECONDARY OUTCOMES:
: Quality of life questionnaire that measures the patients' physical and psychological well-being. | Pre-procedure measurement and another measurement will be assessed one month after first procedure
  Health related quality of life questionnaire its simplified (HRQOL S36) will be used to quantify degree of improvement of physical and psychological well being.The questionnaire is formed of 8 domains,each domain is scaled from 0-100,0 is the worst disability and 100 is the best .Patient is said to be improved when improvemnt of 30% baseline take place

CONTACTS AND LOCATIONS:
Locations (1):
- maha sadek El Derh, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided